CLINICAL TRIAL: NCT05955651
Title: Prospective Analysis to Detect Myometrial Cells in Peritoneal Washing in Patients Undergoing Minimally Invasive Hysterectomy Using Containment Bag at University of Texas Medical Branch
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0269
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; Pelvic washings; Myometrial cell spillage; Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic washings: Three Samples of peritoneal washings will be collected and send to pathology. looking for myometrial cell spillage at three designated points in surgery. 1st before hysterectomy, 2nd after hysterectomy, and 3rd after morcellation and extraction of the uterus out of the abdominal cavity.
  Interventions: Diagnostic Test: Peritoneal washings

INTERVENTIONS:
Diagnostic Test: Peritoneal washings — Peritoneal washing will be done at designated point in the surgical procedure. one hundred cc of normal saline, will be used to irrigate the peritoneal cavity. Samples of the fluid will be collected, with the goal to collect as much fluid as possible for the study, with minimum of 60 cc should be collected. Samples will be sent to the pathology lab.
  1. First washing will be collected after obtaining entry into the peritoneal cavity with placement of the first laparoscopic trocar, before any manipulation of the uterus.
  2. Second washing will be done after the hysterectomy and containment of the uterus in the bag.
  3. Third washing will be collected after scalpel morcellation of the uterus in the containment bag, extraction and closure of the vaginal cuff.

SUMMARY:
The Aim of the study is to determine endometrial/myometrial spillage during total laparoscopic hysterectomy with manual morcellation.

DETAILED DESCRIPTION:
This will be a single institution prospective analysis study. The study will include 50 women who are undergoing minimally invasive hysterectomy. Surgery will be done from 08/01/2023 to 08/01/2024, for benign conditions with uterus that is > 10 cm that requires contained bag morcellation such as (Fibroids, Adenomyosis, Endometriosis, abnormal uterine bleeding, pelvic organ prolapse). Three Samples of peritoneal washings will be collected and send to pathology. First washing will be collected after entering the abdominal cavity, second washing will be done after completion of hysterectomy and containment of the uterus in the bag, and the third washing after scalpel morcellation of the uterus in the containment bag and extraction within the bag. Extraction of the specimen will be done either through the vagina or through a mini laparotomy incision (2-3 cm).

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing minimally invasive Laparoscopic / Robotic hysterectomy for presumably benign conditions such as (fibroids, adenomyosis, endometriosis, pelvic organ prolapse, abnormal uterine bleeding)
2. Large size uterus measuring more than 10 cm on US requiring cold knife morcellation within the Alexis containment bag, surgery will be done by designated surgeon at UTMB from 08/01/2023 to 08/01/2024.
3. Women 18 years and older
4. Subjects must be able to provide consents.
5. Normal endometrial biopsy.
6. Normal cervical cancer screening

Exclusion Criteria:

1. Known Gynecological malignancy.
2. Endometrial biopsy with endometrial intraepithelial hyperplasia.
3. History of exposure to pelvic radiation
4. Post-menopausal patients
5. Emergency hysterectomy
6. TDC patients
7. Patient less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women needing minimally invasive hysterectomy for benign conditions, 18 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Detection of myometrial cell spillage in peritoneal washing | Pelvic washing samples will be sent the pathology lab to be examined within 2 days of the surgery.
  To evaluate potential cell spillage from morcellated tissue, the 3 peritoneal washings collected will be sent to cytology lab to be examined for the presence of smooth muscle cells

SECONDARY OUTCOMES:
Timing of myometrial cell spillage during hysterectomy | Pelvic washing samples will be sent the pathology lab to be examined within 2 days of the surgery.
  To determine at what stage myometrial cell spillage happens during a minimally invasive hysterectomy surgery (before, after completion of the hysterectomy or after morcellation and tissue extraction)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No